CLINICAL TRIAL: NCT01801423
Title: Primary Prevention of Strokes in Nigerian Children With Sickle Cell Disease Affiliated Titles: Sickle Cell Disease - Stroke Prevention in Nigeria (SPIN) Trial
Brief Title: Sickle Cell Disease - Stroke Prevention in Nigeria Trial
Acronym: SPIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Aminu Kano Teaching Hospital (Other)
Responsible Party: Principal Investigator, Michael DeBaun, Vice Chair for Clinical Research, JC Peterson Endowed Chair, Professor of Pediatrics and Medicine, Director, Vanderbilt-Meharry-Matthew Walker Center of Excellence in Sickle Cell Disease, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R01NS094041-01 (NIH); 1R01NS094041-01 (NIH); 1R21NS080639-01 (NIH)
Record Dates: First submitted 2013-02-26; First posted 2013-02-28 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Sickle Cell Anemia; Sickle Cell Disease; Stroke
Keywords: transcranial Doppler; stroke; sickle cell anemia; Nigeria; hydroxyurea; low income country
MeSH Terms: conditions — Anemia, Sickle Cell; Stroke | interventions — Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hydroxyurea (Experimental): Study investigators propose to enroll 60 children with SCA and an elevated TCD measurement between 5 and 12 years of age in this one arm feasibility study of hydroxyurea therapy, with follow-up of at least 12 months per subject. The study intervention will include HU to begin at ~ 20 mg/kg/day(range 17.5 - 26 mg/kg/day). No dose escalation will occur. Given the success of the first year of enrollment and the favorable response of TCD measurement after 3 months on HU therapy, the study investigators have participants as an internal pilot. The definitive phase III trial will now compare low dose HU therapy to the result of no treatment arm from the STOP Trial.
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea — Hydroxyurea will be prescribed as an investigational therapy by the treating physician. Recommended guidelines for titration of hydroxyurea to maximal tolerated dose are below. The study intervention will include hydroxyurea to begin at ~20 mg/kg/day (range 17.5 - 26 mg/kg/day). No dose escalation will occur as this dose was shown to have some efficacy in infants with SCA and was associated with rare myelosuppression.(1)
  Other Names: Droxia; Hydrea; Mylocel

SUMMARY:
Given large absolute numbers of individuals with sickle cell disease in Nigeria, hydroxyurea therapy for all individuals with sickle cell disease may not be initially feasible; however, a targeted strategy of hydroxyurea use for primary prevention of strokes is an alternative to the standard therapy (observation) for high-risk individuals. The investigators propose a feasibility study, Sickle Cell Disease - Stroke Prevention in Nigeria (SPIN) Trial, to determine whether hydroxyurea can be used for primary prevention of strokes in Nigerian children with sickle cell anemia.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is the most common genetic disease in the world. Approximately 150,000 Nigerian children are born each year with SCD, making it the country with the largest burden of sickle cell disease in the world. SCD is the most common cause of stroke in children and results in considerable morbidity in affected children. The current primary prevention approach of regular monthly blood transfusion therapy of children at high risk of stroke (identified by elevated transcranial Doppler measurements) is not feasible in a low income country such as Nigeria due to scarcity of supply, cost, and high rate of blood borne infections. In the United States, hydroxyurea (HU) is standard therapy for adults with SCD and may be a reasonable prevention alternative to regular blood transfusion for treatment of primary stroke in high-risk children. Given large absolute numbers of individuals with SCD in Nigeria, HU therapy for all individuals with SCD may not be initially feasible; however, a targeted strategy of HU use for primary prevention of strokes is an alternative to the standard therapy (observation) for high-risk individuals. Study investigators therefore propose a feasibility study to determine the acceptability of HU for primary prevention of strokes in Nigerian children with sickle cell anemia (SCA) in preparation for a National Institute of Health (NIH) sponsored Phase III Trial. Investigators will establish a safety protocol for using HU in a clinical trial setting and complete the necessary preparations for a definitive phase III trial. To accomplish these aims study investigators have assembled a strong multidisciplinary team representing Vanderbilt University and two premier in-country institutions: Aminu Kano Teaching Hospital, Nigeria, and Friends in Global Health-Nigeria. Completion of a definitive trial will not only benefit children with SCA in sub-Saharan Africa, where the majority of children with SCA live in the world, but could provide reasonable evidence for an alternative to blood transfusion therapy for the primary prevention of strokes in the US. To our knowledge this would be the first stroke prevention trial in Nigeria and could establish a precedent to expand to secondary stroke prevention for children and adults with SCA, as regrettably, no therapy is available to prevent recurrent stroke in these high-risk patients in resource-poor nations.

ELIGIBILITY:
Inclusion Criteria for Screening:

* Patients with hemoglobin SS or S beta zero thalassemia confirmed by hemoglobin electrophoresis;
* Informed consent from a parent or legal guardian and assent of participant ages 5 through 12;
* Successful completion of screening procedures: cerebral blood flow velocity ≥ 200 cm/sec in the terminal portion of the middle cerebral artery;
* Patient must be 5 through 12 years of age (i.e., must have attained their 5th but not their 13th birthday when the consent is signed).

Exclusion Criteria for Screening:

* Prior overt stroke (a focal neurological deficit of acute onset) by history, focal neurological deficit on standardized neurological examination, or concern for moderate or severe neurological deficit (which could be due to stroke) based on a positive "10 questions" screening (an established tool in resource poor countries).(2,3) A "positive" screening is defined as answering yes to any one of the 10 questions. The negative predictive value (child does not have moderate or several neurological impairment) of the "10 questions" is greater than 94% in children (2);
* Other exclusions: significant cytopenias [absolute neutrophil count (ANC) <1500/ul, platelets <150,000/ul, reticulocytes <80,000/ul, unless Hb is > 9 g/dl], renal insufficiency (creatinine > 0.8 mg/dl); other significant organ system dysfunction, or other contraindication to hydroxyurea therapy; and history of seizures or diagnosis of epilepsy;
* Patients for whom hydroxyurea therapy is under consideration prior to study consent/education;
* Patients who have previously been treated with hydroxyurea and are being considered to restart hydroxyurea therapy;
* Other significant organ system dysfunction;
* Any other condition or chronic illness, which in the opinion of the site's Principal Investigator (PI) makes participation ill-advised or unsafe.
* Participants of child bearing age who are pregnant or may become pregnant should not take hydroxyurea. If a participant becomes pregnant during the study, their hydroxyurea treatment will be stopped immediately. The onsite will notify the clinical coordinating center and the principal investigators of the case. The site principal investigator and study principal investigators will determine what therapy the participant should receive during pregnancy that is of standard care.

Inclusion Criteria for Study Therapy:

* Successful completion of screening procedures inclusive of cerebral blood flow velocity greater than or equal to 200 cm/sec measured twice or at least one measurement greater than or equal to 220 cm/sec in the terminal portion of the middle cerebral artery or two TCD measurements above 190 cm/sec within a three month interval;
* Informed consent from a parent or legal guardian for study therapy and assent of the participant completed;
* Participant is able to swallow a capsule as observed by study personnel;
* Acceptance of hydroxyurea therapy for one year. After one year of therapy, the participant will have the option to continue therapy with follow up visits to monitor adherence to therapy.

Exclusion Criteria for Treatment Group:

- Unable to commit to follow up visits for the course of the study.

Inclusion Criteria for participants that are not eligible to receive hydroxyurea therapy, but will be followed for one year (control group):

* Successful completion of screening procedures inclusive of cerebral blood flow velocity less than or equal to 199 cm/sec in the terminal portion of the middle cerebral artery;
* Informed consent from a parent or legal guardian and assent from the participant;
* Acceptance to be followed for one year in the study. Hydroxyurea may be given for other reasons as part of the participant's ongoing care, but it will not be given as part of the study.

Exclusion Criteria for the treatment and control groups:

- Unable to commit to follow up visits for the course of the study.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2013-04-24 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Hydroxyurea Therapy Acceptance and Adherence | 5 years
  The primary outcome measure will be adherence to daily administration of hydroxyurea. If adherence rate is less than 55%, alternative strategies must be considered for the definitive Phase III Trial.

SECONDARY OUTCOMES:
Hydroxyurea Safety protocol for Children with Sickle Cell Anemia | 12 Months
  Study investigators will evaluate the use of a standard safety protocol, non-dose escalating, for hydroxyurea in children with sickle cell anemia using a protocol similar to the recently completed National Heart Lung and Blood Institute (NHLBI) Baby HUG study, published in Lancet.(1) Study investigators expect the proportion of serious adverse reactions, as well as hydroxyurea-related morbidity and mortality, to be very small compared to the benefits. Study investigators will compare the frequency of severe adverse events and hydroxyurea toxicity related events that are associated with hospitalization in those receiving hydroxyurea (n= 60) to those who had normal transcranial Doppler measurements (n= 210) over the course of one year.

OTHER OUTCOMES:
Feasibility of a Definitive Phase III Trial for Hydroxyurea Therapy to Prevent Strokes in Sickle Cell Disease | 24 Months
  During the course of the current study, study investigators will prepare a manual of operations and case report forms for the proposed trial. Investigators will also solidify working relationships with our colleagues and collaborators at Aminu Kano Teaching Hospital in Kano, Nigeria; and develop and organize all committees, collaborators and study procedures necessary for initiation of a successful, definitive, Phase III Trial.

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. DeBaun, MD, MPH, Principal Investigator — Vanderbilt University; Muktar Aliyu, MBBS, MPH, DrPH, Principal Investigator — Vanderbilt University; Lori Jordan, MD, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Aminu Kano Teaching Hospital, Kano, Nigeria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang WC, Ware RE, Miller ST, Iyer RV, Casella JF, Minniti CP, Rana S, Thornburg CD, Rogers ZR, Kalpatthi RV, Barredo JC, Brown RC, Sarnaik SA, Howard TH, Wynn LW, Kutlar A, Armstrong FD, Files BA, Goldsmith JC, Waclawiw MA, Huang X, Thompson BW; BABY HUG investigators. Hydroxycarbamide in very young children with sickle-cell anaemia: a multicentre, randomised, controlled trial (BABY HUG). Lancet. 2011 May 14;377(9778):1663-72. doi: 10.1016/S0140-6736(11)60355-3. PMID 21571150
- [Background] Mung'ala-Odera V, Meehan R, Njuguna P, Mturi N, Alcock K, Carter JA, Newton CR. Validity and reliability of the 'Ten Questions' questionnaire for detecting moderate to severe neurological impairment in children aged 6-9 years in rural Kenya. Neuroepidemiology. 2004 Jan-Apr;23(1-2):67-72. doi: 10.1159/000073977. PMID 14739570
- [Background] Mung'ala-Odera V, Newton CR. Identifying children with neurological impairment and disability in resource-poor countries. Child Care Health Dev. 2007 May;33(3):249-56. doi: 10.1111/j.1365-2214.2006.00714.x. PMID 17439437